CLINICAL TRIAL: NCT04674956
Title: A Prospective, Randomized, Double-blinded, Multi-center Clinical Trial to Evaluate the Efficiency and Safety of Anti-PD1 Antibody (Camrelizumab) Combined With Paclitaxel(Albumin Bound) and Gemcitabine Versus Paclitaxel(Albumin Bound) and Gemcitabine as First-line Therapy in Patients With Metastatic Pancreatic Cancer
Brief Title: A Prospective, Randomized, Double-blinded, Multi-center Clinical Trial to Evaluate the Efficiency and Safety of Anti-PD1 Antibody (Camrelizumab) Combined With Paclitaxel(Albumin Bound) and Gemcitabine as First-line Therapy in Patients With Metastatic Pancreatic Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, liwei wang, Director of department of oncology, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPOG1210-07
Record Dates: First submitted 2020-12-15; First posted 2020-12-19 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Cancer Stage IV; Pancreatic Cancer Metastatic
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — camrelizumab; Taxes; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Patients are assigned into 2 arms randomly of 1：1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participant and investigators are masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): Regimens：anti-PD1 antibody and AG regimens.
  Interventions: Drug: Camrelizumab; Drug: Paclitaxel(Albumin Bound) and Gemcitabine
- Control arm (Placebo Comparator): Regimens：Placebo and AG regimens.
  Interventions: Drug: Paclitaxel(Albumin Bound) and Gemcitabine; Drug: Placebo

INTERVENTIONS:
Drug: Camrelizumab — PD-1 antibody（Camrelizumab）, 200mg, D1; every 21 days as a cycle.
  Arms: Treatment arm
Drug: Paclitaxel(Albumin Bound) and Gemcitabine — Paclitaxel(Albumin Bound), 125 mg/m2D18; Gemcitabine, 1000mg/m2D1, 8;every 21 days as a cycle.
Drug: Placebo — Placebo, 200mg, D1; every 21 days as a cycle.
  Arms: Control arm

SUMMARY:
Aim：Evaluate the efficiency and safety of anti-PD1 antibody (Camrelizumab) combined with Paclitaxel(Albumin Bound) and Gemcitabine as first-line therapy in patients with metastatic pancreatic cancer.

Drug information：

* anti-PD1 antibody (Camrelizumab)
* AG regimens：the standard first-line regimens for metastatic pancreatic cancer.

DETAILED DESCRIPTION:
CPOG1210-07 is a prospective, randomized, double-blinded, multi-center clinical trial in China aiming to evaluate the efficiency and safety of anti-PD1 antibody (Camrelizumab) combined with Paclitaxel(Albumin Bound) and Gemcitabine versus Paclitaxel(Albumin Bound) and Gemcitabine as first-line therapy in patients with metastatic pancreatic cancer.

The anti-PD1 antibody(Camrelizumab) is a humanized monoclonal antibody which can specifically bind to PD-1 and block the interaction between PD-1 and its ligand (PD-L1), allowing T cells to recover the immune response against tumors. It is proved to be effective in certain cancers such as ovarian cancers and certification proved by Chinese Food and Drug Administration(CFDA) includes Hodgkin's lymphoma, non-small cell lung cancer, esophageal cancer and liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged >= 18 years, male or female; 2. Histologically or Cytologically confirmed metastatic pancreatic adenocarcinoma; 3. Patients have never received systematical anti-cancer therapy; 4. Based on Response Evaluation Criteria In Solid Tumors (RECIST1.1), there should be at least one measurable lesion which has never received local treatment like radiotherapy(The lesion located in previous radiotherapy areas can also be selected as target lesions if the progress confirmed.) 5. ECOG:0-1; 6. Expected survival>=12 weeks; 7. Essential organs function must meet the following criteria (Any blood products, growth factor, leucocyte promoting drugs, platelet promoting drugs, drugs for anemia are not allowed in 14 days before the first use of the experimental medication):

  1. Absolute neutrophil count(ANC) >= 1.5x10^9/L
  2. Platelet >= 85x10^9/L
  3. Hemoglobin >= 90g/L
  4. Serum Albumin >= 30g/L
  5. Total bilirubin <= 2.0 ULN (Biliary obstructive patients after biliary drainage <= 2.5 ULN), AST and ALT <= 3.0 ULN (patients with liver metastasis <= 5 ULN);
  6. Creatinine clearance rate >60 mL/min;
  7. Activated Partial Thromboplastin Time and International Standardized Ratio <= 1.5 ULN (Patients using stable dose of anticoagulant therapy such as low molecular weight heparin or warfarin and INR is within the expected range of anticoagulants can be selected.)

Exclusion Criteria:

* 1. Patients with central nervous system metastasis. 2. Patients only have local advanced diseases. 3. Patients have uncontrolled pleural, pericardial or abdominal effusion requiring drainage.

  4. Patients with history of allergy to monoclonal antibodies, any component of SHR-1210, paclitaxel(Albumin Bound) and Gemcitabine.

  5. Patients have ever received anti PD-1 or anti PD-L1 therapy in the past. 6. Patients have accepted any experimental medication.within 4 weeks before the first dose of our experimental medication administration.

  7. Patients are enrolled in another clinical trial except for observational clinical trial (Non-interventional) or the follow-up of the interventional clinical trial. 8. Patients accepted the last dose of anti-cancer therapy (including radiotherapy) within 4 weeks before the first dose of experimental medication administration.

  9. Patients who need corticosteroid or other immunosuppressive agents. 10. Patients who ever received anti-cancer vaccine or have received live vaccine within 4 weeks before the first dose of administration.

  11. Patients who have received major surgery within 4 weeks before the first dose of administration.

  12. Patients with active autoimmune diseases, history of autoimmune diseases. 13. History of immunodeficiency, including HIV positive test, or other acquired, congenital immunodeficiency disorders, or history of organ transplantation and allogeneic bone marrow transplantation.

  14. Patients with uncontrolled cardiovascular clinical symptoms or diseases. 15. Severe infections occurred within 4 weeks before the first administration. 16. History of interstitial lung disease and non- infectious pneumonia. 17. Patients with active pulmonary tuberculosis (APTB) infection confirmed by medical history or CT examination.

  18. Patients with active hepatitis B or hepatitis C. 19. Patients with any other malignant tumors diagnosed within 5 years before the first administration.

  20. Pregnant or lactating women. 21. According to the researchers, participants have other factors that may force them to end up the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progress free survival | 3 years
  Time until progress free since randomized.

SECONDARY OUTCOMES:
Objective Response Rate | 3 years
  Rate of participants with complete response and partial response.
Disease Control Rate | 3 years
  Rate of participants with complete response and partial response and stable disease.
Duration of Response | 2 years
  Time until progress（PD） since first evaluation as CR or PR.

OTHER OUTCOMES:
CA19-9 in serum | 3 years
  CA19-9 in serum

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Ruijin hospital, Shanghai, Shanghai Municipality
  - Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Renji hospital, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided
Share within six months after the trial complete. IPD: Study protocol，statistical analysis plan，informed consent form and clinical study report.